CLINICAL TRIAL: NCT05796011
Title: PET-CT-based Study of Central Mechanisms of Cortical Metabolism in 18F-FDG and 18F-AV1451 Age-related Deafness: a Cross-sectional Study
Brief Title: PET-CT-based Study of Central Mechanisms of Cortical Metabolism in 18F-FDG and 18F-AV1451 Age-related Deafness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-139-01
Record Dates: First submitted 2023-03-08; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-02

CONDITIONS: Age-related Hearing Loss; PET-CT
Keywords: PET-CT; Age-related hearing loss; 18F-FDG; 18F-AV1451; Cortical metabolism
MeSH Terms: conditions — Presbycusis | interventions — Hearing Aids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Age-related hearing loss patients with hearing aid(s): Age-related hearing loss patients who were fitted with at least one hearing aid.
  Interventions: Device: hearing aids
- Age-related hearing loss patients without an hearing aid: Age-related hearing loss patients who were treated without hearing intervention.
  Interventions: Other: without hearing intervention
- Elderly healthy control: healthy elderly with normal hearing tested by pure tone audiometry.
  Interventions: Other: healthy control

INTERVENTIONS:
Device: hearing aids — Hearing aid(s) fitted for one or two sides of ear.
  Groups: Age-related hearing loss patients with hearing aid(s)
Other: without hearing intervention — neither earing aids nor other heaing treatment were applied.
  Groups: Age-related hearing loss patients without an hearing aid
Other: healthy control — healthy control
  Groups: Elderly healthy control

SUMMARY:
The participants were recruited from elderly subjects in the age range of 60-85 years and audiological assessments, cognitive function assessments, non-invasive brain imaging, behavioral assessments were collected from the normal control group, the elderly deaf non-hearing group and the elderly deaf hearing group according to the inclusion and exclusion criteria. The project aims to investigate the differences in auditory speech and cognitive function in age-related deafness at the behavioural level, and to investigate the central cortical metabolic mechanisms in age-related deafness at the brain imaging level.

DETAILED DESCRIPTION:
The participants were recruited from elderly subjects in the age range of 60-85 years and audiological assessments (pure tone audiometry, speech audiometry), cognitive function assessments (Simple Mental State Examination MMSE scale, Montreal Cognitive Assessment Scale MoCA scale), non-invasive brain imaging (functional near-infrared spectroscopy fNIRS, EEG/ERP), behavioral assessments (functional near-infrared spectroscopy fNIRS, EEG/ERP, PET/CT, etc.) were collected from the normal control group, the elderly deaf non-hearing group and the elderly deaf hearing group according to the inclusion and exclusion criteria. The project aims to investigate the differences in auditory speech and cognitive function in age-related deafness at the behavioural level, and to investigate the central cortical metabolic mechanisms in age-related deafness at the brain imaging level.

ELIGIBILITY:
Inclusion Criteria:

* age>50yrs，≤85yrs；
* Normal control group: normal hearing, no MCI, i.e. mean air conduction hearing threshold (0.5, 1, 2, 4 kHz) < 25 dB HL, no air-bone conduction difference, MMSE score of 27-30; MoCA (corrected for educational attainment) score of 26-30;
* Elderly deafness without hearing aid group: patients diagnosed with elderly deafness, i.e. as a symmetrical, slowly progressive, binaural occurrence with age. hearing loss and reduced speech recognition with predominantly high frequency hearing involvement in the first place, with reference to the Expert Consensus on the Diagnosis and Intervention of Hearing Loss in the Elderly 2019 edition, mean air conduction threshold (PTA) > 25 dB HL, mean air conduction hearing threshold at high frequency (HF-PTA) > 25 dB HL, no poor air bone conduction, and no previous hearing aid use.
* No major neurological disorders, serious systemic diseases, family history of genetic predisposition, major psychological disorders.

Exclusion Criteria:

* Pure tone audiometric cues with an average pure tone hearing threshold (500Hz, 1kHz, 2kHz, 4kHz) > 91dB HL.
* Excluding diseases such as noise deafness and drug-induced deafness.
* Basic information is incomplete.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants recruited were elderly subjects in the age range of 60-85 years, and normal controls, elderly deaf non-hearing aid group were collected according to the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
pure tone average | through study completion, an average of 6 months
  The pure tone hearing threshold of each octave was tested under standard test conditions. Pure tone average(PTA, an average air conductance threshold of 500, 1000, 2000 and 4000Hz) and high frequence pure tone average(HF-PTA, an average air conductance threshold of 2000, 4000 and 8000Hz) were calculated for analysis
Speech recognition score | through study completion, an average of 6 months
  Speech recognition score was tested under standard test conditions.The stimulus material is a two-syllable word list of Mandarin speech audiometry materials.
MMSE score and grade | through study completion, an average of 6 months
  The scale is divided into seven aspects, including time orientation, place orientation, immediate memory, attention and gauging, delayed memory, language and visual space. There are 30 items in the scale, with a total score of 30. Normal 27 to 30, mild cognitive impairment 21 to 26, moderate cognitive impairment 10 to 20, and severe cognitive impairment 0 to 9.
MoCA score and grade | through study completion, an average of 6 months
  Montreal Cognitive Assessment (Montreal Cognitive Assessment) is a rapid screening tool for abnormal cognitive function. The scoring criteria were: 26 to 30 points for normal cognitive impairment, 18 to 25 points for mild cognitive impairment, 10 to 17 points for moderate cognitive impairment, and 0 to 9 points for severe cognitive impairment.
Otorhinolaryngological diseases and daily life self-assessment questionnaire | through study completion, an average of 6 months
  The questionnaire included otitis media, tinnitus, deafness, ear pain, ear tightness, ear leakage, ear itching, course of disease, severity of self-complaint, etc
Resting Electroencephalogram | through study completion, an average of 6 months
  Electroencephalogram (EEG) is applied to collect the spontaneous and rhythmic biologic potential data of the subjects' resting brain, namely, 8-minute resting state data with their eyes closed without any visual or auditory stimulation, in a dark environment.
Functional Near-Infrared Spectoscopy | through study completion, an average of 6 months
  Functional near-infrared Spectoscopy(fNIRS) is used to collect the changes of oxygenated hemoglobin and deoxygenated hemoglobin in the temporal lobe of a subject during brain activity by using a portable Near Infrared optical signal analysis system from Shimadsu, Japan.
Positron emmision tomography | through study completion, an average of 6 months
  Pet-ct, Positron emmision tomography is adopted by Siemens PET/CT integrated machine in Germany.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided